CLINICAL TRIAL: NCT06697340
Title: The Effect of the Braden Pressure Ulcer Scale on the Prediction of Intensive Care Unit Length of Stay
Brief Title: Braden Pressure Ulcer Scale for Prediction of the Intensive Care Length of Stay
Acronym: BRILS
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cihangir Doğu, Associate Professor, Ankara City Hospital Bilkent
Other Study IDs: TABED 2-24-618
Record Dates: First submitted 2024-11-15; First posted 2024-11-20 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-01

CONDITIONS: Intensive Care Unit ICU; Length of ICU Stay; Pressure Ulcer Risk; Scale Reliability Validity
Keywords: Braden risk assesment scale; Length of stay; ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group I: Intensive Care patients admitted to tertiary intensive care unit and treated more than 24 hours

SUMMARY:
The aim of this study is to predict the length of intensive care unit stay of patients treated in a tertiary general intensive care unit with the help of the Braden risk assesment scale, which is used to predict the risk of pressure ulcers. The main question it aims to answer is:

* Does high Braden scales predict the long lenght of stay? Braden scales of patients admitted to the intensive care unit were recorded every day.

DETAILED DESCRIPTION:
Intensive care units are specialized units where patients with multiple comorbidities are treated. The length of stay in intensive care varies according to the characteristics of the patient, the disease and the center. Prolonged intensive care stay causes an increase in mortality . It has been reported that the severity of the disease as well as the comorbidities of the patients contribute to prolonged stay . One third of patients with stay longer than seven days were evaluated as more fragile than before hospital admission. Prolonged intensive care length of stay leads to an increase in morbidity and mortality, bed demand and costs.

The Braden pressure ulcer scale was developed by Braden et al. in 1987 . Scoring is done under six different headings evaluating sensory perception, humidity, activity, mobility, nutrition and friction/cutting. It has been reported as an effective tool for evaluating pressure ulcer development in intensive care patients. In this scoring system, there are different assessment steps such as mobility, nutrition, sensory perception, etc., which allows the assessment of the functional capacity of the patients at the time of admission. In a study of elderly dementia patients, the Braden scale was found to be effective in predicting 90-day mortality. In a retrospective evaluation of patients with heart failure, the Braden scale was reported to predict 30-day mortality.

The aim of our study is to predict the length of intensive care stay by analyzing the Braden scales calculated on the day of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients treated in intensive care
* Patients treated with diagnoses other than Covid-19
* Patients without missing data in the hospital electronic data system
* Patients hospitalized for more than 24 hours

Exclusion Criteria:

* Patients younger than 18 years
* Patients treated for Covid-19 disease
* Patients with missing data in the hospital electronic data system
* Patients hospitalized for less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical and surgical intensive care patients admitted to the tertiary general intensive care unit of Ankara Bilkent City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Intensive care length of stay | Time period between patient admission to intensive care unit and patient discharge, patient transfer to ward or patient death, whichever came first. Estimated time up to 52 weeks
  Patient intensive care length of stay

SECONDARY OUTCOMES:
Mortality | Time interval between patient intensive care unit admission to patient mortality. Estimated time is up to 52 weeks
  All-cause mortality rate in the intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng H, Ling Y, Li Q, Tang Y, Li X, Liang X, Huang X, Su L, Lyu J. ICU admission Braden score independently predicts delirium in critically ill patients with ischemic stroke. Intensive Crit Care Nurs. 2024 Jun;82:103626. doi: 10.1016/j.iccn.2024.103626. Epub 2024 Jan 13. PMID 38219301
- [Background] Cheng H, Li X, Liang X, Tang Y, Wei F, Wang Z, Lyu J, Wang Y. Braden score can independently predict 90-day mortality in critically ill patients with dementia. Int J Geriatr Psychiatry. 2024 May;39(5):e6093. doi: 10.1002/gps.6093. PMID 38752607
- [Background] Bandle B, Ward K, Min SJ, Drake C, McIlvennan CK, Kao D, Wald HL. Can Braden Score Predict Outcomes for Hospitalized Heart Failure Patients? J Am Geriatr Soc. 2017 Jun;65(6):1328-1332. doi: 10.1111/jgs.14801. Epub 2017 Feb 21. PMID 28221672